CLINICAL TRIAL: NCT00269191
Title: A 12-Week, Randomized, Placebo- and Active-Comparator-Controlled, Parallel-Group, Double-Blind Study to Assess the Safety and Efficacy of Etoricoxib 30 mg Versus Ibuprofen 2400 mg in Patients With Osteoarthritis (Study 1)
Brief Title: A Study to Assess the Safety and Efficacy of an Investigational Drug in Patients With Osteoarthritis (0663-071)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-071; 2005_110
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
Keywords: Arcoxia
MeSH Terms: conditions — Osteoarthritis | interventions — Etoricoxib; Duration of Therapy; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, etoricoxib / Duration of Treatment 12 Weeks
Drug: Placebo or Ibuprofen / Duration of Treatment 12 Weeks

SUMMARY:
This study was conducted to assess the safety and tolerability of the drug and to evaluate its efficacy in the treatment of osteoarthritis of the hip or knee in men and women.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical and radiographic diagnosis of osteoarthritis of the hip or knee
* Either prior NSAID or Acetaminophen users within the the ARA functional class I,II or III
* Patients required to demonstrate a "flare" of the signs and symptoms of OA following withdrawal of NSAID treatment
* Prior acetaminophen users also required to demonstrate greater than a defined minimum level of signs and symptoms of OA.

Exclusion Criteria:

* No history of concurrent arthritic disease
* uncontrolled hypertension or an active cardiac condition
* No history of hepatitis, neoplastic disease, stroke or transient ischemic attack within a specified duration.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2003-02-05 (Actual); Primary Completion 2003-11-07 (Actual); Study Completion 2003-11-21 (Actual)

PRIMARY OUTCOMES:
Pain and physical function over 12-weeks as assessed by the WOMAC VA 3.0 pain subscale, WOMAC VA 3.0 physical function subscale, and Patient Global Assessment of Disease Status, as well as safety over 12-weeks as assessed by adverse experiences.

SECONDARY OUTCOMES:
Patient Global Assessment of Response to Therapy, Investigator Global Assessment of Disease Status, Stiffness, and Overall WOMAC scales as assessed over 12-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Wiesenhutter CW, Boice JA, Ko A, Sheldon EA, Murphy FT, Wittmer BA, Aversano ML, Reicin AS; Protocol 071 Study Group. Evaluation of the comparative efficacy of etoricoxib and ibuprofen for treatment of patients with osteoarthritis: A randomized, double-blind, placebo-controlled trial. Mayo Clin Proc. 2005 Apr;80(4):470-9. doi: 10.4065/80.4.470. PMID 15819283
- [Background] Laine L, Curtis SP, Cryer B, Kaur A, Cannon CP; MEDAL Steering Committee. Assessment of upper gastrointestinal safety of etoricoxib and diclofenac in patients with osteoarthritis and rheumatoid arthritis in the Multinational Etoricoxib and Diclofenac Arthritis Long-term (MEDAL) programme: a randomised comparison. Lancet. 2007 Feb 10;369(9560):465-73. doi: 10.1016/S0140-6736(07)60234-7. PMID 17292766